CLINICAL TRIAL: NCT04068402
Title: Optimization of the Vivio System Algorithm as an Aid in the Identification of Heart Sounds Associated With Severe Aortic Stenosis
Brief Title: Vivio AS (Aortic Stenosis) Algorithm Optimization Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company changed strategic direction in Oct 2019
Sponsor: Avicena LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VS-001-AO
Record Dates: First submitted 2019-07-25; First posted 2019-08-28 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-01

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Masking Description: No masking required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Vivio System

INTERVENTIONS:
Device: Vivio System — The Vivio System is an electronic auscultatory device and optical sensor, plus software application intended to provide support to the physician in the evaluation of heart sounds in patients. The product will analyze the acoustic signals of the heart and signals from a captured arterial (carotid) waveform. The analysis procedure will identify and analyze specific heart sounds and arterial waveform features captured by the Vivio device, to devise a scoring system for severe aortic stenosis.

SUMMARY:
Optimize a candidate software algorithm using data collected with the Vivio system for use as an aid in the identification of heart sounds associated with severe aortic stenosis

DETAILED DESCRIPTION:
Prospective, non-randomized, single-center study of adult subjects referred for echocardiography. Total of 200 enrolled subjects at 1 site

Enrolled subjects will undergo:

Vivio system data capture, standard of care transthoracic echocardiogram (TTE). Vivio analysis will not be available to non-Avicena personnel

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (21 years of age or older).
2. Referred for transthoracic echocardiography by physician/primary care provider/cardiologist.
3. Willing and able to participate in all study evaluations and allow access to medical testing and records.
4. Ability to understand and sign an informed consent or have a legally authorized representative to provide informed consent on behalf of the subject.

Exclusion Criteria:

1. Acute coronary syndrome, cardiogenic shock or the need for inotropic/mechanical circulatory support.
2. Need for bedside echocardiogram (inpatient).
3. Prosthetic device previously implanted at aortic valve position.
4. Inability to palpate carotid pulse
5. History of carotid sinus hypersensitivity (i.e. fainting in response to touching or positioning the neck).
6. History of significant carotid artery disease or treatment (surgery, stenting, > 50% stenosis in both left and right carotid artery).
7. Open skin lesions at target site of Vivio examination.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint - Generation of an optimized algorithm that can be used to develop an algorithm for use as an aid in the identification of heart sounds associated with severe aortic stenosis. | 48 hours
  Generation of an optimized algorithm that can be used to develop an algorithm for use as an aid in the identification of heart sounds associated with severe aortic stenosis.

SECONDARY OUTCOMES:
Secondary Endpoint - Incidence of Adverse Events: Summary of all reported adverse events during the study | 48 hours
  Incidence of Adverse Events: Summary of all reported adverse events during the study. Events will be summarized by seriousness (e.g. serious vs. non-serious), attribution (e.g. device vs. procedure vs. comorbidity) based upon site reported data.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Brady, JD, Study Director — Avicena LLC
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States